CLINICAL TRIAL: NCT07003737
Title: Short-term Blinatumomab Intensification for MRD-Negative Acute B-Cell Lymphoblastic Leukemia Before Allogeneic Hematopoietic Stem Cell Transplantation: A Prospective, Multicenter, Randomized Controlled Study
Brief Title: Blinatumomab Intensification for MRD-Negative Acute B-Cell Lymphoblastic Leukemia Before Allogeneic Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yanmin Zhao, Vice Director, Bone Marrow Transplantation Center, the First Affiliated Hospital, School of Medicine, Zhejiang University, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLI4MRD-BALL
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphoblastic Leukemia, B-precursor
Keywords: allogeneic hematopoietic stem cell transplantation; measurable residual disease; Blinatumomab; high-risk BCR::ABL1-negative
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — blinatumomab; Consolidation Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Non-BiTE group) (Sham Comparator): Patients proceed directly to allo-HSCT without blinatumomab intensification.
  Interventions: Other: Consolidation Chemotherapy or Direct Allogeneic HSCT
- Blinatumomab Group (BiTE group) (Experimental): Patients receive short-term blinatumomab intensification before undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT).
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab is administered starting approximately one month before allogeneic hematopoietic stem cell transplantation (allo-HSCT).
  For participants weighing ≥45 kg: 9 μg/day is administered on Days 1-3, followed by 28 μg/day on Days 4-14.
  For participants weighing <45 kg: 5 μg/m²/day (based on body surface area) is administered on Days 1-3, followed by 15 μg/m²/day on Days 4-14. The total dose must not exceed the dosage used for participants ≥45 kg.
  Arms: Blinatumomab Group (BiTE group)
Other: Consolidation Chemotherapy or Direct Allogeneic HSCT — Participants in the Non-BiTE group will either proceed directly to allogeneic hematopoietic stem cell transplantation (allo-HSCT) or receive one additional cycle of consolidation chemotherapy prior to
  Arms: Control Group (Non-BiTE group)

SUMMARY:
This is a prospective, multicenter, randomized controlled trial designed to evaluate whether short-term blinatumomab intensification before allogeneic hematopoietic stem cell transplantation (allo-HSCT) can improve survival outcomes in adults with high-risk BCR::ABL1-negative B-cell acute lymphoblastic leukemia (B-ALL) who have achieved measurable residual disease (MRD) negativity. Blinatumomab, a CD19/CD3 bispecific T-cell engager, has shown promising efficacy in eradicating MRD and prolonging survival in B-ALL patients. In this study, eligible participants will be randomly assigned to receive either short-term blinatumomab consolidation prior to allo-HSCT or proceed directly to allo-HSCT. The primary endpoint is relapse-free survival (RFS). This study aims to optimize treatment strategies and improve long-term outcomes for patients with high-risk BCR::ABL1-negative B-ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with B-cell acute lymphoblastic leukemia (B-ALL) according to the 2022 WHO classification.

2. Age between 18 and 65 years. 3. Meets the National Comprehensive Cancer Network (NCCN) criteria for high-risk B-ALL, based on clinical or cytogenetic/molecular features:

1. Clinical high-risk features (any of the following):

   1. Age > 35 years
   2. Peripheral WBC count > 30 × 10⁹/L
   3. Cytogenetic/molecular high-risk features (any of the following):
2. Cytogenetic and molecular high-risk features (at least one of the following):

   1. Hypodiploidy (<44 chromosomes)
   2. TP53 mutation
   3. KMT2A rearrangement
   4. MLL rearrangement
   5. HLF rearrangement
   6. ZNF384 rearrangement
   7. MEF2D rearrangement
   8. MYC rearrangement
   9. BCR-ABL1-like (Ph-like) ALL, including:
   10. JAK pathway rearrangements (CRLF2r, EPORr, JAK1/2/3r, TYK2r, SH2B3 mutation, IL7R mutation, JAK1/2/3 mutations)
   11. ABL-class rearrangements (ABL1, ABL2, PDGFRA, PDGFRB, FGFR1)
   12. Other kinase fusions (e.g., NTRK3r, FLT3r, LYNr, PTK2Br)
   13. PAX5alt
   14. t(9;22)(q34.1;q11.2); BCR-ABL1 with IKZF1 mutation and/or prior chronic myeloid leukemia (CML)
   15. Intrachromosomal amplification of chromosome 21 (iAMP21)
   16. IKZF1 alteration
   17. Complex karyotype (≥5 chromosomal abnormalities) 4. CD19-positive by immunophenotyping. 5. BCR::ABL1-negative. 6. Achieved complete remission (CR) after induction therapy. 7. Measurable residual disease (MRD)-negative by flow cytometry (FCM). 8. Availability of a matched sibling donor, haploidentical related donor, or matched/unmatched unrelated donor.

       9. ECOG performance status score of 0-2. 10. Creatinine clearance ≥ 60 mL/min (by Cockcroft-Gault formula). 11. AST and ALT ≤ 3 × upper limit of normal (ULN); total bilirubin ≤ 2 × ULN. 12. Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiography. 13. Expected survival > 8 weeks. 14. Signed written informed consent, with ability to understand and comply with the study protocol.

       Exclusion Criteria:
       1. Prior exposure to blinatumomab, chimeric antigen receptor (CAR) T-cell therapy, or anti-CD22 immunotoxins.
       2. Clinically significant cardiovascular disease, including uncontrolled arrhythmia, uncontrolled hypertension, congestive heart failure, NYHA class III or IV heart disease, or myocardial infarction within 3 months prior to screening.
       3. Other severe comorbidities that may limit participation in the trial (e.g., severe infection, renal failure).
       4. Known HIV infection or uncontrolled severe viral hepatitis.
       5. Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2028-02-05 (Estimated)

PRIMARY OUTCOMES:
2-year Relapse-Free Survival (RFS) | 2 years after transplantation
  Relapse-free survival is defined as the time from transplantation to either disease relapse or death from any cause, whichever occurs first. Patients who are alive and relapse-free at 2 years will be considered as having achieved 2-year RFS.

SECONDARY OUTCOMES:
Cumulative Incidence of Relapse (CIR) | Up to 2 years after transplantation
  Defined as the cumulative incidence of hematologic relapse, accounting for competing risks such as non-relapse mortality.
Non-Relapse Mortality (NRM) | Up to 2 years after transplantation
  Death from any cause without prior hematologic relapse.
Incidence of Hematologic and Non-Hematologic Adverse Events | From first dose of study drug to 100 days post-transplant
  Safety evaluation based on CTCAE v5.0 criteria, including treatment-related cytopenias, infections, neurotoxicity, and other adverse events.
Measurable Residual Disease (MRD) Status | From enrollment to up to 2 years after transplantation
  MRD status assessed using multi-parameter flow cytometry or PCR prior to HSCT. Evaluated as MRD-negative or MRD-positive.
2-year Overall Survival (OS) | 2 years after transplantation
  Overall survival is defined as the time from HSCT to death from any cause. Patients alive at 2 years are considered to have achieved 2-year OS.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided